CLINICAL TRIAL: NCT00601497
Title: Effects of Electrical Stimulation on Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Ann Gill Taylor, RN, EdD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIC 11630
Record Dates: First submitted 2008-01-12; First posted 2008-01-28 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: InterX 5000
- 2 (Placebo Comparator)
  Interventions: Device: InterX 5000

INTERVENTIONS:
Device: InterX 5000 — 20-30 minute device sessions on the following schedule: 3 times per week for 3 weeks, then 2 times per week for 3 weeks, then 1 time per week for 2 weeks.
  Other Names: Noninvasive Interactive Neurostimulation

SUMMARY:
The purpose of this study is to find out whether electrical stimulation can reduce knee pain and increase function in people with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Diagnosis of primary osteoarthritis of the knee (as defined by American College of Rheumatology criteria)
* Knee pain of at least six months duration
* Moderate or greater knee pain (defined as a score of 3 or greater on an 11 point numeric pain rating scale) for most days in the last month
* Willing to abide by protocol and treatment schedule.

Exclusion Criteria:

* Implants, such as pacemaker, TENS, or insulin pump, incompatible with electrical stimulation
* Uncontrolled concomitant disease affecting the knee, such as: rheumatoid arthritis, systemic lupus erythema, psoriatic arthritis
* Pregnant or breast-feeding
* Intra-articular corticosteroid or hyaluronic acid injection into the knee within 3 months preceding study
* Arthroscopy of the knee within the past year
* Significant injury to the knee within the past 6 months
* Use of assistive devices other than a cane or knee brace
* Disease of spine or other lower extremity joints of sufficient degree to affect assessment of the knee

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Knee Pain | Baseline, Week 4, Week 8, and Week 12

SECONDARY OUTCOMES:
Knee function | Baseline, Week 4, Week 8, and Week 12
Knee stiffness | Baseline, Week 4, Week 8, and Week 12
Patient global assessment | Baseline, Week 4, Week 8, and Week 12
Health-related quality of life | Baseline, Week 4, Week 8, and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ann G Taylor, RN, EdD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States